CLINICAL TRIAL: NCT03429075
Title: Psilocybin vs Escitalopram for Major Depressive Disorder: Comparative Mechanisms
Acronym: Psilodep-RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Alexander Mosely Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17HH3790; 2017-000219-18 (EudraCT Number)
Record Dates: First submitted 2017-12-06; First posted 2018-02-12 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorder, Major
Keywords: depression; mdd; major depression; major depressive disorder; unipolar depression; psilocybin; psychedelics; psychedelic; escitalopram; ssri
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Psilocybin; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Patients receive Psilocybin
  Interventions: Drug: Psilocybin + Placebo
- Escitalopram (Active Comparator): Patients receive Escitalopram
  Interventions: Drug: Psilocybin + Escitalopram

INTERVENTIONS:
Drug: Psilocybin + Placebo — Multiple dosing days psilocybin vs 6 weeks of daily placebo
  Arms: Psilocybin
Drug: Psilocybin + Escitalopram — Multiple dosing days psilocybin vs 6 weeks of daily escitalopram
  Arms: Escitalopram

SUMMARY:
This is a randomised double-blind clinical trial. The aim is to compare the efficacy and mechanisms of action of psilocybin, the primary psychoactive substance in 'magic mushrooms', with the selective serotonin reuptake inhibitor (SSRI) escitalopram for major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

1. Major depressive disorder (DSM-IV)
2. Depression of moderate to severe degree (17+ on the 17-item Hamilton Depression Scale (HAM-D)).
3. No Magnetic Resonance Imaging (MRI) contraindications
4. No SSRI contraindications
5. Has a general practitioner (GP) or other mental healthcare professional who can confirm diagnosis
6. 18-80 years of age
7. Males and females
8. Sufficiently competent with English language

Key exclusion criteria:

1. Current or previously diagnosed psychotic disorder
2. Immediate family member with a diagnosed psychotic disorder
3. Medically significant condition rendering unsuitability for the study (e.g., diabetes, epilepsy, severe cardiovascular disease, hepatic or renal failure e.g. creatine clearance:renal clearance (CLRC) < 30 ml/min etc.)
4. History of serious suicide attempts requiring hospitalisation.
5. Significant history of mania (determined by study psychiatrist and medical records)
6. Psychiatric condition judged to be incompatible with establishment of rapport with therapy team and/or safe exposure to psilocybin, e.g. borderline personality disorder
7. Blood or needle phobia
8. Positive pregnancy test at screening or during the study, women who are planning a pregnancy and/or women who are nursing/breastfeeding.
9. Participants who do not agree to use an acceptable contraceptive method throughout their participation in study.
10. Current drug or alcohol dependence
11. No email access
12. Use of contraindicated medication
13. Patients presenting with abnormal QT interval prolongation at screening or with a history of this (QTc at screening above 440ms for men and above 470ms for women)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Nutt, Medicine, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carhart-Harris RL, Bolstridge M, Day CMJ, Rucker J, Watts R, Erritzoe DE, Kaelen M, Giribaldi B, Bloomfield M, Pilling S, Rickard JA, Forbes B, Feilding A, Taylor D, Curran HV, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: six-month follow-up. Psychopharmacology (Berl). 2018 Feb;235(2):399-408. doi: 10.1007/s00213-017-4771-x. Epub 2017 Nov 8. PMID 29119217
- [Result] Carhart-Harris R, Giribaldi B, Watts R, Baker-Jones M, Murphy-Beiner A, Murphy R, Martell J, Blemings A, Erritzoe D, Nutt DJ. Trial of Psilocybin versus Escitalopram for Depression. N Engl J Med. 2021 Apr 15;384(15):1402-1411. doi: 10.1056/NEJMoa2032994. PMID 33852780
- [Derived] Erritzoe D, Barba T, Greenway KT, Murphy R, Martell J, Giribaldi B, Timmermann C, Murphy-Beiner A, Jones MB, Nutt D, Weiss B, Carhart-Harris R. Effect of psilocybin versus escitalopram on depression symptom severity in patients with moderate-to-severe major depressive disorder: observational 6-month follow-up of a phase 2, double-blind, randomised, controlled trial. EClinicalMedicine. 2024 Sep 21;76:102799. doi: 10.1016/j.eclinm.2024.102799. eCollection 2024 Oct. PMID 39764567
- [Derived] Peill J, Marguilho M, Erritzoe D, Barba T, Greenway KT, Rosas F, Timmermann C, Carhart-Harris R. Psychedelics and the 'inner healer': Myth or mechanism? J Psychopharmacol. 2024 May;38(5):417-424. doi: 10.1177/02698811241239206. Epub 2024 Apr 12. PMID 38605658
- [Derived] Szigeti B, Weiss B, Rosas FE, Erritzoe D, Nutt D, Carhart-Harris R. Assessing expectancy and suggestibility in a trial of escitalopram v. psilocybin for depression. Psychol Med. 2024 Jun;54(8):1717-1724. doi: 10.1017/S0033291723003653. Epub 2024 Jan 22. PMID 38247730
- [Derived] Nayak SM, Bari BA, Yaden DB, Spriggs MJ, Rosas FE, Peill JM, Giribaldi B, Erritzoe D, Nutt DJ, Carhart-Harris R. A Bayesian Reanalysis of a Trial of Psilocybin versus Escitalopram for Depression. Psychedelic Med (New Rochelle). 2023 Mar;1(1):18-26. doi: 10.1089/psymed.2022.0002. Epub 2022 Oct 28. PMID 37337526
- [Derived] Murphy R, Kettner H, Zeifman R, Giribaldi B, Kartner L, Martell J, Read T, Murphy-Beiner A, Baker-Jones M, Nutt D, Erritzoe D, Watts R, Carhart-Harris R. Therapeutic Alliance and Rapport Modulate Responses to Psilocybin Assisted Therapy for Depression. Front Pharmacol. 2022 Mar 31;12:788155. doi: 10.3389/fphar.2021.788155. eCollection 2021. PMID 35431912
- [Derived] Daws RE, Timmermann C, Giribaldi B, Sexton JD, Wall MB, Erritzoe D, Roseman L, Nutt D, Carhart-Harris R. Increased global integration in the brain after psilocybin therapy for depression. Nat Med. 2022 Apr;28(4):844-851. doi: 10.1038/s41591-022-01744-z. Epub 2022 Apr 11. PMID 35411074

RESULTS

PARTICIPANT FLOW:
Groups:
- Psilocybin: Patients receive two doses of 25mg psilocybin, 3 weeks apart. After the first dose of 25mg psilocybin, patients start taking one daily placebo tablet every morning for 3 weeks. After their second 25mg psilocybin session, patients start taking two daily placebo tablets for another 3 weeks.
  All tablets are identical and visit procedures are identical otherwise.
- Escitalopram: Patients receive two doses of 1mg psilocybin (considered to be virtually placebo), 3 weeks apart. After the first dose of 1mg psilocybin, patients start taking one daily 10mg escitalopram tablet every morning for 3 weeks. After their second 1mg psilocybin session, patients start taking two daily tablets of escitalopram (10mg each, 20mg in total) for another 3 weeks.
  All tablets are identical and visit procedures are identical otherwise.
Period: Overall Study
Arm/Group | Psilocybin | Escitalopram
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psilocybin | Escitalopram | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (11.7) | 39.1 (9.7) | 41.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 19 | 20 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28 | 24 | 52
  Asian | 1 | 4 | 5
  Mixed Asian + White | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 29 | 59
No previous psilocybin use [Number; unit: participants] | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of the BOLD Signal
Description: Patients were tested with functional magnetic resonance imaging (fMRI) to measure brain brain responses to emotional faces before and after the treatment. The 2 values of BOLD signal (before and after exposure to emotional faces) were used to estimate a percentage value per patient and then these were used to estimated a group percentage change.
Time Frame: Baseline measure vs 6 weeks post 1st psilocybin dosing
Population: The data obtained from an imaging group in the trial, in which functional MRI was used to predict responses to the trial drugs, have not been analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in BOLD signal
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 25 | 21
percentage change in BOLD signal | -0.08 (0.45) | 0.43 (0.62)

2. Primary Outcome: Change in QIDS-16: Quick Inventory of Depressive Symptomatology Self-Rated (QIDS-16)
Description: Change in QIDS-16 (self-rated measure of depressive symptoms). Scale is composed of 16 items that correlate with the 9 Diagnostic Statistical Manual (DSM-IV) symptom criteria for depression. Each response is graded 0-4 (none-severe symptoms). Questions 1-4 concern sleep disturbances, Question 5 addresses sad mood, Questions 6-9 appetite/weight, Question 10 concentration, Question 11 self-criticism, Question 12 suicidal ideation, Question 13 interest, Q14 energy/fatigue and Questions 15-16 psychomotor agitation/retardation. All questions that address the same topic are grouped and only the highest score from each group is summed up together with the other questions in order to produce a total score. Scores can range from 0-27 and depression severity is graded based on the total score in the following way: 1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
  Lower score =better outcome (less depression)
Time Frame: Baseline vs 6 weeks post 1st psilocybin dosing
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 30 | 29
score on a scale | -8 (1) | -6 (1)
Statistical Analysis 1: Comparison: Psilocybin vs Escitalopram; Test type: Equivalence — ANCOVA; p = 0.17, ANCOVA

3. Secondary Outcome: Change in Hamilton Depression Scale (HAMD-17)
Description: HAMD-17: clinician rated Hamilton Depression Scale of depression severity. Range of scores: 0-52: where 0-7 is normal, 8-16 is mild, 17-23 is moderate, >23 is severe.
  A threshold score of 17 is the entry: a score of 17 or higher indicated moderate-severe depression and was a requirement for entry into this trial at the screening point. This baseline does not refer to the screening point, it refers to the HAMD conducted 7-10 days before psilocybin dosing.
  A higher decrease in the HAMD (larger negative change score) is a better outcome.
Time Frame: Change from baseline (7-10 days pre-dosing) to 6 weeks after the first psilocybin dose
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 30 | 29
units on a scale | -10.5 (1) | -5.1 (1)

4. Secondary Outcome: Change in Beck Depression Inventory (BDI-IA)
Description: BDI-IA: patient-rated Beck Depression Inventory, depressive symptomatology scale. Higher score = worse depression. The total score range is 0-63: where 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe
  Higher negative score = greater decrease in depression scores 6 weeks after each treatment arm = better outcome.
Time Frame: Change from baseline (7-10 days pre-dosing) to 6 weeks after the first psilocybin dose
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 30 | 29
units on a scale | -18.4 [-22.6 to -13.8] | -10.8 [-14.3 to -7.3]

5. Secondary Outcome: Change in MADRS
Description: MADRS - Montgomery-Asberg Depression Rating Scale, clinician-rated measure of depression. This scale is clinician-rated and consists of 10 items; each item is rated on a 0-6 scale, resulting in a maximum total score of 60 points, with higher scores indicative of greater depressive symptomology.36 The MADRS scoring instructions indicate that a total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates "mild depression," 20 to 34 indicates "moderate depression," a score of 35 and greater indicates "severe depression," and a total score of 60 or greater indicates "very severe depression."
  A higher decrease in the MADRS (larger negative change score) is a better outcome.
Time Frame: Change from baseline (7-10 days pre-dosing) to 6 weeks after the first psilocybin dose
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 30 | 29
score on a scale | 14.4 (1.7) | -7.2 (1.7)

6. Secondary Outcome: Number of Patients Who "Responded": Quick Inventory of Depressive Symptomatology (QIDS-16) Response at 6 Weeks
Description: Number of patients who "responded" on the QIDS-16 scale (Quick Inventory of Depressive Symptomatology, self-rated). "Response" is defined by a decrease in QIDS score of 50% from baseline.
  Higher number of patients who responded = better outcome for treatment arm.
Time Frame: Change from baseline (7-10 days pre-dosing) to 6 weeks after the first psilocybin dose
Measure: Number; unit: participants
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 30 | 29
participants | 21 | 14

7. Secondary Outcome: Number of Patients Who "Remitted": QIDS-16 Remission Rate
Description: Number of patients who "remitted" on the QIDS-16 scale (Quick Inventory of Depressive Symptomatology, self-rated). "Remission" is defined by having a QIDS score below 5 at the 6 week point = no depression.
  Higher remission rate = better outcome (less depressed patients after treatment)
Time Frame: Change from baseline (7-10 days pre-dosing) to 6 weeks after the first psilocybin dose
Measure: Number; unit: participants
Arm/Group | Psilocybin | Escitalopram
Number analyzed (Participants) | 30 | 29
participants | 17 | 8

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Psilocybin | Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 26/30 | 24/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Psilocybin (N=30) | Escitalopram (N=29)
Headache (Nervous system disorders) | 20 | 15
Nausea (Gastrointestinal disorders) | 8 | 9
Fatigue (General disorders) | 2 | 7
Anxiety (Psychiatric disorders) | 0 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 4
Migraine (Nervous system disorders) | 3 | 1
Palpitations (Cardiac disorders) | 1 | 3
Sleep disorder (Psychiatric disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Feeling abnormal (General disorders) | 0 | 3
Feeling jittery (General disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03429075/Prot_000.pdf